CLINICAL TRIAL: NCT06418334
Title: Ultrasonographic Measurement of Diaphragmatic Thickness in Adolescents With Thoracal Hyperkyphosis
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 109
Record Dates: First submitted 2024-01-11; First posted 2024-05-17 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hyperkyphosis; Spine Deformity; Diaphragm Issues
Keywords: Thoracal Hyperkyphosis; Diaphragma Thickness; Ultrasonographic Measurement
MeSH Terms: conditions — Kyphosis | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 10-18 years who were diagnosed with thoracal hyperkyphosis deformity: Thoracal Hyperkyphosis study form consisting of clinical and radiological measurements of patients aged 10-18 years who were diagnosed with thoracal hyperkyphosis deformity and applied to the scoliosis outpatient clinicwill be filled in detail.
  Interventions: Diagnostic Test: Thoracal hyperkyphosis study form; Diagnostic Test: Scoliosis graphy; Diagnostic Test: Pulmonary function test; Diagnostic Test: Ultrasonographic Measurement

INTERVENTIONS:
Diagnostic Test: Thoracal hyperkyphosis study form — Thoracal hyperkyphosis study form consisting of clinical and radiological measurements of patients aged 10-18 years who applied to the outpatient clinic with chest deformity will be filled in detail.
Diagnostic Test: Scoliosis graphy — Patients whose forward bending test and clinical evaluation results are compatible with hyperkyphosis and scoliosis radiographs are requested. Coronal, sagittal balance; coronal and sagittal Cobb angles will be measured from posterior-anterior (PA) and lateral scoliosis radiographs.
Diagnostic Test: Pulmonary function test — Pulmonary function tests (PFTs) are noninvasive tests that show how well the lungs are working. The tests measure lung volume, capacity, rates of flow, and gas exchange. This information can help participant healthcare provider diagnose and decide the treatment of certain lung disorders.
  The investigators will use handheld spirometry device for measurement. Three measurements will be made. In these three measurements; FEV1(Forced Expiratory Volume In One Second)(L), FEV1 (%predicted), FVC (Forced Vital Capacity) (L), FVC (%predicted), FEV1/FVC (%) and FEV1/FVC (%predicted) will be evaluated. The arithmetic average of the results of these three measurements will be taken.
  Other Names: Spirometry Function Test
Diagnostic Test: Ultrasonographic Measurement — Diaphragm thickness will be measured in the supine position with a 6-14 Mhz lineer, conventional ultrasound probe (Mindray DC-8, Shenzen Mindray Bio-Medical Electronics CO. LTD.,P.R. China) at the end of inspiration and expiration from the intercostal space on the anterior axillary line. The measurements will be evaluated by making three measurements from the right 8-9. intercostal space where the diaphragm is best visualized. End-expiratory (Forced residual capacity-FRC) (centimeter-cm), end-inspiratory (Total Lung Capacity) (centimeter-cm) and thickening rate (%) (thickness TLC / thickness FRC) will be evaluated three times and the arithmetic average of these three measurements will be taken.

SUMMARY:
Spinal deformity is common in childhood and adolescence. Any spinal deformity, especially one that affects the thoracic spine, can affect lung function.The diaphragm is the main respiratory muscle, and diaphragm contraction is associated with respiratory functions. The investigators aimed to measure the diaphragmatic thickness in adolescents with increased thoracal kyphosis (thoracal hyperkyphosis) deformities.

DETAILED DESCRIPTION:
Spinal deformity is common in childhood and adolescence, and can often present as scoliosis or increased thoracal kyphosis deformity with various etiologies.

Any spinal deformity, especially one that affects the thoracic spine, can affect lung function. If left untreated, the curves may distort over time as skeletal growth accelerates. In some patients, this can lead to restrictive or obstructive lung disease and, rarely, death as a result of cor pulmonale.

The alignment of the skeletal system in the chest and its harmony with the compliance of the chest wall are related to respiratory function; Thoracic kyphosis and the resulting changes in the rib cage lead to a decrease in lung capacity. The diaphragm is the main respiratory muscle, and diaphragm contraction is associated with respiratory functions. In recent years, ultrasonography (USG) has gained increasing utility for visualizing the diaphragm and assessing its function, with several advantages.

Based on this, the investigators aimed to measure the diaphragmatic thickness in adolescents with increased thoracal kyphosis (thoracal hyperkyphosis) deformities, to show whether there is any relationship between increased kyphosis deformity and diaphragmatic thickness, and to show whether there is any change in diaphragmatic thickness before or after the treatment for kyphosis.

ELIGIBILITY:
Inclusion Criteria:

* Increased thoracal kyphosis (thoracic hyperkyphosis)
* Being between the ages of 10-18

Exclusion Criteria:

* Congenital spinal, costal and diaphragmatic anomalies
* Neuromuscular disease
* Respiratory system diseases that affect lung functions
* Patients who cannot cooperate with spirometry.
* Having surgery to the chest wall or spine

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: It will consist of participants with thoracal hyperkyphosis deformity who apply to the Physical Medicine and Rehabilitation Clinic of the University of Health Sciences Gaziosmanpaşa Training and Research Hospital within the study date ranges, meet the inclusion and exclusion criteria and voluntarily agree to participate in the research. Healthy individuals identical in age and gender will be included in the study as a control group. Demographic information of all individuals involved in the recruitment will be collected.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Thoracal hyperkyphosis study form | Within 1 month of applying to the outpatient clinic
  Thoracal hyperkyphosis study form consisting of clinical and radiological measurements of patients aged 8-18 years who applied to the outpatient clinic with chest deformity will be filled in detail. Coronal, sagittal balance; coronal and sagittal Cobb angles (degree) (degree between upper end vertebral line of thoracal 3 'T3' and lower end vertebral line of 'T12') will be measured from posterior-anterior (PA) and lateral scoliosis radiographs.
Pulmonary function test | Within 1 month of applying to the outpatient clinic
  The investigators will use handheld spirometry device for measurement. Three measurements will be made. In these three measurements; FEV1(Forced Expiratory Volume In One Second) (Liter-L), FEV1 (%predicted) (percentage), FVC (Forced Vital Capacity) (Liter-L), FVC (%predicted) (percentage), FEV1/FVC (%) and FEV1/FVC (%predicted) (percentage) will be evaluated. The arithmetic average of the results of these three measurements will be taken.
Ultrasonographic Measurement | Within 1 month of applying to the outpatient clinic
  Diaphragm thickness (centimeter-cm) will be measured in the supine position with a 6-14 Mhz lineer, conventional ultrasound probe (Mindray DC-8, Shenzen Mindray Bio-Medical Electronics CO. LTD.,P.R. China) at the end of inspiration and expiration from the intercostal space on the anterior axillary line. The measurements will be evaluated by making three measurements from the right 8-9. intercostal space where the diaphragm is best visualized. End-expiratory (Forced residual capacity-FRC) (centimeter-cm), end-inspiratory (Total Lung Capacity) (centimeter-cm) and thickening rate (%) (thickness TLC / thickness FRC) will be evaluated three times and the arithmetic average of these three measurements will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Guneser Gulec, MD, Study Chair — Gaziosmanpasa Training and Research Hospital Physical Rehabilitation Department; Cansu Ozkan, MD, Study Chair — Medical Park Bahcelievler Hospital Physical Medicine and Rehabilitation Department
Locations (1):
- Deniz Oke, Istanbul, Gaziosmanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available on request from the corresponding author (EG). The data will not be publicly available due to their containing information that could compromise the privacy of research participants.

REFERENCES:
- [Result] Jagger F, Tsirikos AI, Blacklock S, Urquhart DS. Adaptation to reduced lung function in children and young people with spinal deformity. J Clin Orthop Trauma. 2020 Mar-Apr;11(2):191-195. doi: 10.1016/j.jcot.2019.12.013. Epub 2020 Jan 3. PMID 32099278
- [Result] Karaali E, Ciloglu O, Gorgulu FF, Ekiz T. Ultrasonographic measurement of diaphragm thickness in patients with severe thoracic scoliosis. J Ultrasound. 2021 Mar;24(1):75-79. doi: 10.1007/s40477-020-00536-w. Epub 2021 Feb 7. PMID 33550575
- [Result] Wang JS. Effect of joint mobilization and stretching on respiratory function and spinal movement in very severe COPD with thoracic kyphosis. J Phys Ther Sci. 2015 Oct;27(10):3329-31. doi: 10.1589/jpts.27.3329. Epub 2015 Oct 30. PMID 26644703
- [Derived] Oke D, Karakullukcuoglu Z, Gulec MG, Ozkan C. Ultrasonographic evaluation of diaphragmatic thickness in adolescents with thoracic hyperkyphosis: new horizons in diagnosis. BMC Musculoskelet Disord. 2026 Jan 2;27(1):92. doi: 10.1186/s12891-025-09462-6. PMID 41484972